CLINICAL TRIAL: NCT05953766
Title: A Randomized Controlled Trial (RCT) Comparing Presacral Nerve Block Versus Sham Block on Post-operative Pain in Women Undergoing Total Laparoscopic Hysterectomy.
Brief Title: Presacral Nerve Block Versus Sham Block on Post-operative Pain for Total Laparoscopic Hysterectomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REB# 21-0104-A
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Post-operative Pain
Keywords: Hysterectomy; Presacral nerve block; Laparoscopy; Anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: We will create a randomization list using a computer-generated allocation sequence in equal ratio with study numbers 1 to 60.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgeon, research team, participants and data analysts will be blinded to treatment group. Our clinic nurse, who works 5 days per week in our ambulatory office and who will have no other role in this study, will prepare the active and placebo syringes and label the syringes according to the randomization list. Each syringe will be prepared individually and provided to the surgeon on the day of surgery. Study participants will be randomized on the day of surgery. The surgeon will instill the drug/placebo from the labeled syringe into the presacral space as the first step prior to starting the hysterectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Presacral Nerve Block (Experimental): Presacral nerve block using 20mL of local ropivacaine 5.0mg/ml instilled in the presacral space
  Interventions: Drug: Ropivacaine injection
- Sham Block (Sham Comparator): 20mL of normal saline (sham block) instilled in the presacral space
  Interventions: Drug: Normal saline injection

INTERVENTIONS:
Drug: Ropivacaine injection — Presacral nerve block using 20mL of local ropivacaine 5.0mg/ml
  Other Names: Naropin
  Arms: Presacral Nerve Block
Drug: Normal saline injection — Sham block using 20 mL of normal saline (0.9% sodium chloride)
  Other Names: Sham block; 0.9% Sodium Chloride
  Arms: Sham Block

SUMMARY:
The study is a single-center parallel group randomized controlled trial comparing the administration of a presacral nerve block using 20mL of local ropivacaine 5.0mg/ml versus 20mL of normal saline (sham block) on post-operative pain following total laparoscopic hysterectomy.

DETAILED DESCRIPTION:
The proposed study is a single-center parallel-group RCT comparing the administration of a presacral nerve block using 20mL of local ropivacaine (5.0mg/ml) versus 20mL of normal saline (sham block). This drug/dose was selected based on the recent study by Rapp et al., which instilled 20mL of ropivacaine into the presacral nerve at the time of open hysterectomy.

Participants will be selected using a convenience sample from Mount Sinai Hospital's outpatient gynecology clinics. All patients age 18 years and older undergoing total laparoscopic hysterectomy will be considered for inclusion. Exclusion criteria include: previous presacral neurectomy, concurrent surgical procedure other than salpingectomy and/or oophorectomy, gynecological cancer beyond stage 1 disease, chronic opioid consumption, fibromyalgia, BMI > 50, language barriers, inability to communicate, or inability to provide consent. All potentially eligible patients will be invited to participate in this study by their surgeon. Interested patients will then meet with a member of the research team to explain the study and obtain informed consent.

The investigators will create a randomization list using a computer-generated allocation sequence in equal ratio (1:1) to either study group with study numbers 1 to 60. A clinic nurse, unaffiliated with any other aspects of the study, who works 5 days per week in the ambulatory office and who will have no other role in this study, will prepare and label the active and placebo syringes according to the randomization list. Each syringe will be prepared individually and provided to the surgeon on the day of surgery.

Study participants will be randomized on the day of surgery. The surgeon will instill the contents from the labeled syringe (either drug/placebo) into the presacral space as the first step prior to starting the hysterectomy.

The surgeon, research team, participants, and data analysts will be blinded to treatment group.

Each study patient will receive standard of care standardized perioperative care as follows:

All patients will receive preoperative multimodal analgesia with acetaminophen 1000 mg.

A protocolized general anesthetic will be used for all patients. Induction of anesthesia will be performed with fentanyl (1-3 mcg/kg), propofol (2-3 mg/kg), and rocuronium (0.6 mg/kg), followed by endotracheal intubation. Patients will be maintained with Sevoflurane anesthetic titrated to a minimum alveolar concentration (MAC) of 0.9-1.2 in a mixture of 50:50 air/oxygen.

Analgesia will be provided with intravenous fentanyl and/or hydromorphone administered to maintain mean arterial pressure or heart rate within 20% of baseline measurements.

At skin closure, unless contraindicated, all patients will be administered intravenously ondansetron 4 mg and IV dexamethasone 0.1 mg/kg for nausea prophylaxis. Unless contraindicated, all patients will also receive intravenous ketorolac 30 mg for analgesia.

Local anesthetic will be provided at the site of the port incisions (2ml per port site of 0.25% bupivacaine with epinephrine).

Following completion of surgery, neuromuscular blockade will be antagonized with neostigmine and glycopyrrolate, and patients will be extubated and brought to the post anesthesia care unit (PACU). As per protocol and routine care, the only adjunctive analgesic administered intra-operatively in addition to opioids will be intravenous ketorolac.

Post-operative pain scores will be assessed using a self-administered numeric rating scale (NRS) for pain at 1, 2 and 3 hours after arrival in the PACU. Those patients with pain scores greater than 4/10 will receive analgesia according to a standard postoperative analgesic regimen. This will consist of intravenous fentanyl 25-50 mcg boluses every 5-10 minutes, intravenous administration of hydromorphone 0.2-0.4 mg boluses as required, and oral administration of either hydromorphone IR 1-2 mg or oxycodone IR 5-10 mg.

Rescue antiemetics will be administered if required at the discretion of the anesthesiologist in the form of IV metoclopramide 5-10 mg, ondansetron 4 mg, or dimenhydrinate 25-50 mg.

Patients will be contacted post-operatively days 1, 2 and 7 in order to collect data on post-operative pain scores, total opioid consumption, and any adverse events (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing total laparoscopic hysterectomy

Exclusion Criteria:

* Previous presacral neurectomy
* Concurrent surgical procedure other than salpingectomy and/or oophorectomy
* Gynecological cancer beyond stage 1 disease
* BMI > 50
* Chronic opioid consumption
* Fibromyalgia
* Language barrier
* Inability to communicate and provide consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-24 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Early post-operative pain at 3 hours following surgery | 3 hours following surgery
  Early post-operative pain measured at 3-hours following surgery by a self-administered numeric pain rating scale (NRS) on a scale from 0 to 10, with 0 indicating no pain and 10 indicating the worst pain imaginable

SECONDARY OUTCOMES:
Post-operative pain at other time points | 1 hour, 2 hour, and post-operative days 1, 2 and 7
  Delayed post-operative pain measured by numeric pain rating scale (NRS) scores at 1 hour, 2 hour, and post-operative days 1, 2 and 7 on a scale from 0 to 10, with 0 indicating no pain and 10 indicating the worst pain imaginable

OTHER OUTCOMES:
Post-operative narcotic usage | Post-operative days 1, 2 and 7
  Total narcotics administered from end of surgery until post-operative days 1, 2 and 7 (calculated from the hospital medical records and pill counts from discharge medications to be elicited by phone the day after surgery)
Adverse effects/complication rates | Post-operative days 1, 2 and 7
  Any negative outcome that is self-reported and elicited from a telephone survey

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No